CLINICAL TRIAL: NCT02847078
Title: Effects of a Smart Phone Application in the Secondary Clinical Prevention Management for Chinese Patients After Coronary Intervention Treatment: a Randomized Controlled Trial
Brief Title: Smart Phone Application in the Secondary Clinical Prevention Management for Chinese Patients
Acronym: SPASCPM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment of patients
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XAJTUFH2016; 2016JM8116 (Other Grant/Funding Number: Science and Technology Department of Shaanxi Province, China)
Record Dates: First submitted 2016-07-13; First posted 2016-07-28 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2016-04

CONDITIONS: Coronary Disease
Keywords: Coronary Disease; percutaneous coronary intervention; secondary prevention; smart phone app
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smart phone app (Experimental): The app contains education materials for secondary prevention of coronary artery disease. So patients can access them very easily. The app pushes heath management recommendation information on the timeline after percutaneous coronary intervention, and also provides health care lecture to help patients to improve their secondary prevention. And online or telephone consultation ways are integrated into the App to provide convenience for patients to communicate with health care professionals.
  Interventions: Device: smart phone app
- Control group (Other): Participants allocated to the control group will receive a booklet with general advice on secondary prevention of coronary artery disease.
  Interventions: Device: A guideline booklet

INTERVENTIONS:
Device: smart phone app — App for this study is provided with real time updating educational materials, reminder, and consultation for improving secondary prevention, and the related information is pushed to a patient in chronological order after his or her PCI operation.
  Arms: Smart phone app
Device: A guideline booklet — A guideline booklet with general advice on secondary prevention of coronary artery disease.
  Arms: Control group

SUMMARY:
The purpose of the study is to investigate the effects of smart phone app on the secondary prevention for patients with coronary heart disease post percutaneous coronary intervention.

DETAILED DESCRIPTION:
The secondary prevention for patients with coronary heart disease post percutaneous coronary intervention (PCI) proved associated with a significant reduction in mortality rates and improvement in quality of life. For the limitation of socio-economic conditions, not all patients post PCI are in a position to receive continuous standardized secondary prevention management. Therefore a smart phone app for secondary prevention management post PCI will be installed on patients' smart phones in order to investigate its effects on risk factors control, medication compliance, as well as quality of life and adverse cardiac events in the next six months post discharge. Participants allocated to the control group will receive a booklet with general advice on secondary prevention of coronary heart disease. Patients in app group and control group will be interviewed by telephone at the 2nd week and the 3rd month, and at the 1st month and 6th month they will return our hospital for face to face follow-up and to compliance and medication adjustment, assessment of life quality, risk factors control and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of coronary heart disease and received a PCI treatment.
* Age 18-65 years.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Speech communication barriers.
* Patients with a clear history of allergies to anti-platelet drugs.
* Patients with a clear history of allergies to anti-platelet ᵦ-blockers.
* Patients with a clear history of allergies to statin drugs.
* Patients with a clear history of allergies to antihypertensive drugs.
* Patients with a clear history of allergies to antidiabetic drugs.
* Patients with serious heart failure(better than NYHA class II).
* Patients with cerebral infarction or cerebral hemorrhage.
* Patients with liver dysfunction (AST and ALT> 2 times that of the reference value).
* Patients with kidney dysfunction (creatinine clearance rate< 60ml/min).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | Baseline and 1 and 6 months
  Seatt1e Angina Questionnaire

SECONDARY OUTCOMES:
Change in medication compliance | Baseline and 1 and 6 months
  Percent of prescribed antiplatelet drug，ᵦ-blocker，angiotensin converting enzyme inhibitor，angiotensin II receptor blocker and statins taken during the past 1 and 6 monthers
Change in systolic blood | Baseline and 1 and 6 months
  systolic blood pressure is measured via pressuremercury sphygmomanometer and recored in the unit of mmHg.
Change in diastolic blood pressure | Baseline and 1 and 6 months
  Diastolic blood pressure is measured via pressuremercury sphygmomanometer and recored in the unit of mmHg.
Changes in serum total cholesterol | Baseline and 1 and 6 months
  Serum total cholesterol is measured by automatic biochemistry analyzer and recorded in the unit of mmol/L.
Changes in serum triglyceride | Baseline and 1 and 6 months
  Serum triglyceride is measured by automatic biochemistry analyzer and recorded in the unit of mmol/L.
Changes in serum high-density lipoproteincholesterol | Baseline and 1 and 6 months
  Serum high-density lipoproteincholesterol is measured by automatic biochemistry analyzer and recorded in the unit of mmol/L.
Changes in serum low-density lipoproteincholesterol | Baseline and 1 and 6 months
  Serum low-density lipoproteincholesterol is measured by automatic biochemistry analyzer and recorded in the unit of mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Hu, Master, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bommer WJ. Coronary revascularization: then, now, future trends. Rev Cardiovasc Med. 2014;15(2):176-7. doi: 10.3909/ricm15-2CAACC. No abstract available. PMID 25051135
- [Result] White CJ. The future of interventional cardiology. Catheter Cardiovasc Interv. 2013 Jan 1;81(1):4-5. doi: 10.1002/ccd.24734. No abstract available. PMID 23281080
- [Result] Sim DS, Kim JH, Jeong MH. Differences in Clinical Outcomes Between Patients With ST-Elevation Versus Non-ST-Elevation Acute Myocardial Infarction in Korea. Korean Circ J. 2009 Aug;39(8):297-303. doi: 10.4070/kcj.2009.39.8.297. Epub 2009 Aug 27. PMID 19949634
- [Result] Pocock S, Bueno H, Licour M, Medina J, Zhang L, Annemans L, Danchin N, Huo Y, Van de Werf F. Predictors of one-year mortality at hospital discharge after acute coronary syndromes: A new risk score from the EPICOR (long-tErm follow uP of antithrombotic management patterns In acute CORonary syndrome patients) study. Eur Heart J Acute Cardiovasc Care. 2015 Dec;4(6):509-17. doi: 10.1177/2048872614554198. Epub 2014 Oct 9. PMID 25301783
- [Result] Goel K, Lennon RJ, Tilbury RT, Squires RW, Thomas RJ. Impact of cardiac rehabilitation on mortality and cardiovascular events after percutaneous coronary intervention in the community. Circulation. 2011 May 31;123(21):2344-52. doi: 10.1161/CIRCULATIONAHA.110.983536. Epub 2011 May 16. PMID 21576654
- [Result] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Result] Heo J, Chun M, Lee KY, Oh YT, Noh OK, Park RW. Effects of a smartphone application on breast self-examination: a feasibility study. Healthc Inform Res. 2013 Dec;19(4):250-60. doi: 10.4258/hir.2013.19.4.250. Epub 2013 Dec 31. PMID 24523989
- [Result] Svetkey LP, Batch BC, Lin PH, Intille SS, Corsino L, Tyson CC, Bosworth HB, Grambow SC, Voils C, Loria C, Gallis JA, Schwager J, Bennett GG. Cell phone intervention for you (CITY): A randomized, controlled trial of behavioral weight loss intervention for young adults using mobile technology. Obesity (Silver Spring). 2015 Nov;23(11):2133-41. doi: 10.1002/oby.21226. PMID 26530929